CLINICAL TRIAL: NCT04564443
Title: A Multi-center, Randomized Controlled Clinical Investigation Evaluating a Unique Micro Water Jet Technology Device Versus Standard Debridement in the Treatment of Diabetic Foot
Brief Title: A Unique Micro Water Jet Technology Device Versus Standard Debridement in the Treatment of Diabetic Foot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medaxis, LLC (Industry)
Collaborators: Professional Education and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDX-DT-01
Record Dates: First submitted 2020-09-22; First posted 2020-09-25 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Alginates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (Medaxis Debritom+™) micro fluid jet wound therapy (Experimental): Medaxis Debritom+™ is a high-quality, micro fluid jet therapy device designed to remove fibrin, necrotic tissue, and biofilm from wound surfaces by mechanical cleaning and stimulation of the diabetic foot wound
  Interventions: Other: Medaxis Debritom+; Other: Additional Outer Dressing Application; Other: Offloading; Other: Fibracol Wound Dressing
- Sharp Surgical Debridement (Active Comparator): Use of a surgical scalpel or curette to remove fibrin, necrotic tissue and biofilm from wound surfaces by mechanically cleaning the wound
  Interventions: Other: Sharp Surgical Debridement; Other: Additional Outer Dressing Application; Other: Offloading; Other: Fibracol Wound Dressing

INTERVENTIONS:
Other: Medaxis Debritom+ — Advanced micro fluid jet therapy to clean and stimulate wound
  Arms: (Medaxis Debritom+™) micro fluid jet wound therapy
Other: Sharp Surgical Debridement — Scalpel or Curette to clean and debride wound
  Arms: Sharp Surgical Debridement
Other: Additional Outer Dressing Application — Application of moisture retentive dressing, and a multi layer compression dressing
Other: Offloading — Patient will be offloaded in a diabetic camboot after treatment, or total contact cast if patient cannot be fit with diabetic offloading boot
  Other Names: Pressure Relief
Other: Fibracol Wound Dressing — Application of a collagen alginate dressing
  Other Names: Calcium Alginate

SUMMARY:
The purpose of this clinical investigation is to assess performance of the Medaxis Debritom+™ and to collect subject outcome data in the treatment of diabetic foot ulcers (DFU) vs Standard sharp debridement.

DETAILED DESCRIPTION:
The economic burden of DFUs costs the United States over $50 billion each year. The cost to treat one subject with DFUs ranges from $11,700 to $16,883. Although approximately 70% of DFUs are shown to heal with good SOC, at least 30% become chronic wounds. These non-healing wounds are at greater risk for infection and lower extremity amputation. Consequently, good standard of care therapy is important for subjects with chronic DFUs to improve subject outcomes, lower treatment costs and reduce the risk of complications.

The removal of necrotic tissue such as slough, eschar, and underlying biofilm constitutes one of the most important parts of standard of care (SOC). Currently, a variety of techniques are used to debride chronic wounds, such as larval therapy, autolytic and enzymatic methods, monofilament polyester fiber pads or brushes, and mechanical debridement with curettes and scalpels. It has also been demonstrated that more frequent debridement, on average, results in faster wound healing. While regarded as the "gold standard," sharp debridement requires considerable experience of clinicians to ensure that contaminated and devitalized tissue is entirely removed without extensively damaging surrounding healthy tissue. Moreover, a recent research has demonstrated that even when surgical debridement is well-conducted so that it removes the majority of biofilm, within 72 hours, biofilm often re-establishes itself. Given that perhaps 60% of chronic wounds have been found to harbor biofilm, it is challenging to keep such wounds free of biofilm so that the wound-healing process can be sustained. Consequently, any method that could potentially remove more biofilm and/or prevent its recurrence could improve the wound healing trajectory.

Medaxis Debritom+™ cleans and stimulates acute and chronic wounds precisely in a tissue-preserving manner. Its high-pressure micro fluid jet removes slough such as fibrin, necrosis or biofilm, as well as foreign bodies, in effect providing an efficient irrigation and debridement of contaminated wounds. The purpose of this clinical investigation is to assess performance of Medaxis Debritom+™ and to collect subject outcome data in the treatment of diabetic foot ulcers (DFU) vs Standard sharp debridement.

There are two arms in the study:

Arm 1: The Experimental Arm , that will include SOC Therapy. SOC therapy in this study is offloading of the DFU (CAM boots or total contact casting [TCC] if the subject's foot is too large for a CAM), use of the Medaxis Debritom+™ micro jet to clean the wound followed by a wound care covering ( Fibracol dressing or equivalent) along with a moisture retention dressing and a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll and compression wrap (DynaflexTM or equivalent).

Arm 2: The Standard of Care Arm. The SOC therapy in this study is offloading of the DFU (CAM boots or total contact casting [TCC] if the subject's foot is too large for a CAM), appropriate sharp or surgical debridement, followed by a wound care covering (Fibracol dressing or equivalent) along with a moisture retention dressing and a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll and compression wrap (DynaflexTM or equivalent).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Presence of a diabetic foot ulcer (DFU) meets all of the following features: Wagner Grade 1 or 2 (see Appendix A for definitions), including wounds that extend to the ligament, tendon, joint capsule or fascia
* At least 50% below the medial aspect of the malleolus
* Without abscess or osteomyelitis
* The index ulcer will be the largest ulcer if two or more DFUs are present and will be the only one evaluated in the study. If other ulcerations are present on the same foot, they must be more than 2 cm distant from the index ulcer.
* The index ulcer (i.e. current episode of ulceration) has been present for greater than 4 weeks prior to SV1 and less than 1 year, as of the date the subject consents for study.
* The index ulcer is a minimum of 1.0 cm2 and a maximum of 25 cm2 at SV1 and TV1.
* Adequate circulation to the affected foot as documented by a dorsal transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, or an Ankle Branchial Index (ABI) between 0.7 and 1.3 within 3 months of SV1, using the affected study extremity. As an alternative arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle within 3 months of SV1.
* The index ulcer has been offloaded for at least 14 days prior to randomization.
* Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, IUD's, barriers or abstinence) during the course of the study and undergo pregnancy tests.
* Subject understands and is willing to participate in the clinical study and can comply - with weekly visits.
* Subjects must have read and signed the IRB approved ICF before screening procedures are undertaken.

Exclusion Criteria:

* The index ulcer is deemed by the investigator to be caused by a medical condition other than diabetes.
* The index ulcer, in the opinion of the investigator, is suspicious for cancer or has a positive carcinoma diagnosis.
* Subjects with a history of more than two weeks of treatment with immune-suppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within 1-month prior to first SV1, or who receive such medications during the screening period or who are anticipated to require such medications during the course of the study.
* Subjects taking a selective COX-2 inhibitor, such as Celecoxib, for any condition.
* Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding SV1.
* History of radiation at the ulcer site (regardless of time since last radiation treatment).
* Index ulcer has been previously treated or will need to be treated with any prohibited therapies. (See Section 6.2.4 of this protocol for a list of prohibited medications and therapies).
* Subjects with a previous diagnose of HIV, Hepatitis C, or other contagious diseases
* Presence of any condition(s) which seriously compromises the subject's ability to complete this study or the subject has a known history of poor adherence with medical treatment.
* Osteomyelitis or bone infection of the affected foot as verified by x-ray, CAT Scan, or MRI within 30 days prior to randomization. (In the event of an ambiguous diagnosis, the Principal Investigator will make the final decision).
* Subject is pregnant or breast-feeding.
* Presence of diabetes with poor metabolic control as documented with an HbA1c > 12.0 within 90 days of randomization.
* Subjects with end stage renal disease as evidenced by a serum creatinine ≥ 3.0 mg/dL within 6 months of randomization.
* Index ulcer has reduced in area by 20% or more after 14 days of SOC from SV1 to the TV1/randomization visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of wounds completely healed at or before 16 weeks | 16 weeks
  examine the time it takes the wound to heal over a 16 week period

SECONDARY OUTCOMES:
Incidence of any index wound-related cellulitis or infection by 16 weeks | 16 weeks
  examine the number of subject that develop wound cellulitis or infection over 16 weeks
Cost of treatment, including any index wound-related complications, by 16 weeks | 16 weeks
  examine the cost of all treatments within 16 weeks
Percent Area Reduction at 16 weeks. | 16 weeks
  examine the reduction in wound size at 16 weeks
Cost of hospitalization for any index wound-related event, including any wound recurrence involving the area of the index wound by 16 weeks | 16 weeks
  examine the patient hospitalization costs for wound related event over 16 weeks
Incidence of hospitalization between randomization and EOS for any index wound-related event, including any wound recurrence involving the area of the index wound | 16 weeks
  examine the incidence of subject being hospitalized during the study period
Moleculight imaging | 2 weeks
  Difference in wound bioburden from wound biopsy
Kent Imaging - Snapshot camera | 16 weeks
  test oxygenation of wound tissue

CONTACTS AND LOCATIONS:
Overall Officials: Robert Galiano, MD, Principal Investigator — Northwestern University School of Medicine; David Armstrong, DPM, MD, PhD, Principal Investigator — University of Southern California; Keck School of Medicine
Locations (6):
- United States (6):
  - CCR Research, San Francisco, California
  - Doctors Research Network, South Miami, Florida
  - Foot and Ankle Associates of the Mid-Atlantic, Frederick, Maryland
  - Foot and Ankle Associates of the Mid-Atlantic, Raleigh, North Carolina
  - Lower Extremity Institute for Research and Therapy, LLC, Youngstown, Ohio
  - Foot and Ankle Associates of the Mid-Atlantic, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No